CLINICAL TRIAL: NCT03832868
Title: Evaluating the Impact of Decision Aid Timing on Mandatory Shared Decision Making for Defibrillator Implantation
Brief Title: Syngery-Evaluating the Impact of Decision Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Faisal Merchant MD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00107168
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Implantable Cardioverter-defibrillators (ICDs)
Keywords: Decision aid

STUDY DESIGN:
Intervention Model Description: Clinic sites will be block-randomized to eliminate contamination induced by individual-level randomization for a system-level intervention. Each site will rotate on a monthly basis whether the decision aid is administered pre- or post-office visit, and this will be applied to all ICD patients. Each site will have a minimum of 2 months exposure to each "arm." No blinding will occur.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-visit decision aid (Experimental): Patients receiving the decision aid pre-visit will be given a paper copy of the decision aid in the waiting room and will have a minimum of 15 minutes to review it - either in the waiting room or in the exam room while waiting for the electrophysiologist.
  Interventions: Behavioral: Pre-visit timing of receipt of the ICDs implantation decision aid
- Post-visit decision aid (Experimental): Patients receiving the decision aid after the encounter will meet with the electrophysiologist first and receive the aid afterward.
  Interventions: Behavioral: Post-visit timing of receipt of the ICDs implantation decision aid

INTERVENTIONS:
Behavioral: Pre-visit timing of receipt of the ICDs implantation decision aid — The intervention is the timing of receipt of the decision aid. The decision aid is designed to facilitate informing patients and helping to reach a decision.The implantable cardioverter-defibrillators (ICDs) implantation decision aid presents treatment options, risks, and benefits in lay terms.It is currently utilized in all of the Emory cardiac electrophysiology clinics as part of usual clinical care.
  Arms: Pre-visit decision aid
Behavioral: Post-visit timing of receipt of the ICDs implantation decision aid — The intervention is the timing of receipt of the decision aid. The decision aid is designed to facilitate informing patients and helping to reach a decision.The implantable cardioverter-defibrillators (ICDs) implantation decision aid presents treatment options, risks, and benefits in lay terms.It is currently utilized in all of the Emory cardiac electrophysiology clinics as part of usual clinical care.
  Arms: Post-visit decision aid

SUMMARY:
The aim of this study is to determine whether it is better to give patients an implantable cardioverter-defibrillators (ICDs) decision aid before they have their first consultation with an implanting cardiac electrophysiologist or after the consult.

DETAILED DESCRIPTION:
There are many unanswered questions about how shared decision making should be executed and how decision aids should be employed. The aim of this study is to determine whether it is better to give patients an implantable cardioverter-defibrillators (ICDs) decision aid before they have their first consultation with an implanting cardiac electrophysiologist or after the consult.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* evaluated for primary prevention implantable cardioverter-defibrillators (ICDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Decisional ICDs knowledge score among pre-visit arm participants compare to post-visit arm participants | Date of ICD implantation (up to 60 days from the date of receiving the decision aid)
  Patients will receive a survey including 11 questions to gauge decisional knowledge about ICDs. The survey is expected to take no more than 10-15 minutes to complete, which should allow adequate time for completion in the pre-procedure area without interrupting clinical workflow.

SECONDARY OUTCOMES:
Decision Conflict Scale score among pre-visit arm participants compare to post-visit arm participants | Date of ICD implantation (up to 60 days from the date of receiving the decision aid)
  Patients will receive a survey including 12 questions to measure decisional conflict. The surveys are expected to take no more than 10-15 minutes to complete, which should allow adequate time for completion in the pre-procedure area without interrupting clinical workflow.
Values-choice ICDs concordance score among pre-visit arm participants compare to post-visit arm participants | Date of ICD implantation (up to 60 days from the date of receiving the decision aid)
  Patients will receive a survey including 12 questions to measure values-choice concordance. The surveys are expected to take no more than 10-15 minutes to complete, which should allow adequate time for completion in the pre-procedure area without interrupting clinical workflow.

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Merchant, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Data is being collected in REDCAP and is deidentified. The study team will have the tool to match subjects if needed. The team has no current plans to share data, but can if necessary (including the data dictionaries). All data can be shared after being deidentified.The study team can share the protocol, statistical plan, ICF, and survey tool. The decision tool is already available. Data will be available immediately following publication and for 3 years after. Those requesting access to data should contact the principal investigator (Dr. Faisal Merchant). Requests will be evaluated based on need and data usage agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available immediately following publication and for 3 years after.
Access Criteria: Those requesting access to data should contact the principal investigator (Dr. Faisal Merchant). Requests will be evaluated based on need and data usage agreement.